CLINICAL TRIAL: NCT01621425
Title: Lean Body Mass as a Determinant of Docetaxel Pharmacokinetics and Toxicity
Acronym: LEANDOC
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF 11.01
Record Dates: First submitted 2012-05-25; First posted 2012-06-18 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer; Metastatic Castration-resistant Prostate Carcinoma
Keywords: breast cancer; prostate carcinoma; docetaxel; lean body mass; Body Surface Area; body weight; dexascan
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Body Weight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for docetaxel concentration measurement (n=4)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TAC regimen: Female subject diagnosed with breast carcinoma and will receive docetaxel treatment according to standard hospital protocol
  Interventions: Other: Lean body mass; Other: Total body weight; Other: bloodsampling
- PRODOC regimen: male subject diagnosed with metastatic castration-resistant prostate carcinoma and will receive docetaxel treatment according to standard hospital protocol
  Interventions: Other: Lean body mass; Other: Total body weight; Other: bloodsampling

INTERVENTIONS:
Other: Lean body mass — Lean Body mass (DEXA scan and Bioelectrical Impedance Assessments) within one week prior to the first docetaxel dose
Other: Total body weight — Total Body weight (TBW) (scale) within one week prior to the first docetaxel dose
Other: bloodsampling — Blood samples will be taken during the first docetaxel administration of the first cycle, just before docetaxel infusion (t=0 min.), 30 min after start of infusion (t=30 min.), just prior to end of infusion (t=55 min.) and between 3 to 6 hours post start infusion following a limited sampling model

SUMMARY:
Docetaxel is used as a first line anti-cancer drug in the treatment of several cancers, mainly breast- and metastatic castration-resistant prostate carcinoma.

Anti-cancer drugs are being dosed based on patients estimated Body Surface Area in order to equalize total drug exposure. Nevertheless, docetaxel treatment is characterized by highly interindividual pharmacokinetic variation leading to toxicity and under-treatment.

The investigators will determine which anthropometric parameters, LBM, total body weight (TBW) or BSA correlate best to docetaxel exposure (AUC) for both males and females.

DETAILED DESCRIPTION:
Docetaxel is used as a first line anti-cancer drug in the treatment of several cancers, mainly breast- and metastatic castration-resistant prostate carcinoma.

Anti-cancer drugs are being dosed based on patients estimated Body Surface Area in order to equalize total drug exposure. Nevertheless, docetaxel treatment is characterized by highly interindividual pharmacokinetic variation leading to toxicity and under-treatment.

For most anti-cancer drugs, including docetaxel, other anthropometric parameters, such as Lean Body Mass (LBM), have been suggested to be superior to Body Surface Are (BSA) as a determinant for dosing but this has not been implemented in clinical practice.

The investigators will determine which anthropometric parameters, LBM, total body weight (TBW) or BSA correlate best to docetaxel exposure (AUC) for both males and females.

The investigators will determine if occurrence of docetaxel toxicity can be related to dose/LBM.

The investigators will determine which methods to measure LBM: DEXA, Bioelectrical Impedance Assessments (BIA) or formula estimates are accurate enough for dosing calculations to be used for dosing docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations
* Female subject diagnosed with breast carcinoma and will receive docetaxel treatment according to standard hospital protocol (TAC regimen) or male subject diagnosed with metastatic castration-resistant prostate carcinoma and will receive docetaxel treatment according to standard hospital protocol (PRODOC regimen)
* Subject has a live expectancy of 12 weeks or greater
* Absolute neutrophile count (ANC) > 1.5 x 10E9/L
* Platelet count > 100 x 10E9/L
* Serum creatinine ≤ 2 x ULN
* Total bilirubin level < 1.5 x ULN

Exclusion Criteria:

* Docetaxel treatment within the last year
* Moderate or severe liver impairment; [ALAT and/or ASAT ≥ 1.5 ULN] and [AF ≥ 2.5 ULN]
* Current therapy with any drug, dietary supplements, or other compounds, or have been used in the last 2 weeks prior to the first docetaxel administration, known to inhibit or induce CYP3A4.
* Inability to understand the nature and extent of the study and the procedures required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 female subjects who are diagnosed with breast and 20 male subjects with metas-tatic castration-resistant prostate carcinoma and will receive docetaxel treatment according to standard hospital protocol (TAC or PRODOC regimens)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
anthropometric parameters related to exposure | within one week prior to first docetaxel dose
  To determine which anthropometric parameters, LBM, total body weight (TBW) or BSA correlates best to docetaxel exposure (AUC) for both males and females

SECONDARY OUTCOMES:
relation between docetaxel toxicity and dose/LBM | 1 cycle (21 days)
  can docetaxel toxicity be related to dose/LBM? docetaxel toxicity is defined as: number of rates of grade 3/4 toxicity, dose delay, dose reduction, treatment termination and combinations of all four as Dose-Limiting Toxicity (DLT)
determine the best method to measure lean body mass | within one week prior to first docetaxel dose
  To determine which methods to measure LBM: Bioelectrical Impedance As-sessments (BIA) or formula estimates are accurate enough for dosing calculations to be used for dosing docetaxel. These methods will be compared to the LBM derived from the DEXA scan as the general accepted, accurate and validated method for determining LBM.

CONTACTS AND LOCATIONS:
Overall Officials: Rien Hoge, PharmD, Principal Investigator — Deventer Ziekenhuis; Frank Jansman, PharmD, PhD, Study Chair — Deventer Ziekenhuis
Locations (2):
- Netherlands (2):
  - Deventer Hospital, Deventer
  - Radboud University Nijmegen Medical Centre, Nijmegen